CLINICAL TRIAL: NCT06881147
Title: Effects of Physiotherapy Combined With Botulinum Neurotoxin in Patients With Cervical Dystonia With and Without an Effective Sensory Trick: Clinical and Functional MRI Findings
Brief Title: Physiotherapy and Botox for Cervical Dystonia: Impact of Sensory Tricks and Brain Imaging Insights
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS San Raffaele (Other)
Collaborators: Ospedale San Luca, Istituto Auxologico Italiano, Milano (Unknown)
Responsible Party: Principal Investigator, Prof. Massimo Filippi, MD, IRCCS San Raffaele
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: DYT_sensory_trick
Record Dates: First submitted 2025-02-11; First posted 2025-03-18 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Cervical Dystonia
MeSH Terms: conditions — Torticollis

STUDY DESIGN:
Intervention Model Description: It is a comparative study: two parallel groups will undergo the same treatment. Patients will be included if they have a Cervical Dystonia both with and without and effective sensory trick. The recruited patients will be divided into two groups according to the presence of an effective sensory trick (DYT-trick and DYT-no-trick groups).
Who Masked: Outcomes Assessor
Masking Description: The statistician will be blind about the characteristics of the two groups. Considering the different clinical phenotypes of patients (DYT-trick and DYT-no-trick) clinical evaluators and physiotherapists cannot be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Patients with Cervical Dystonia and an effective sensory trick (DYT-trick) (Experimental): Patients with an effective sensory trick will undergo a multimodal physiotherapy program for 6 weeks
  Interventions: Behavioral: Multimodal physiotherapy program
- Patients with Cervical Dystonia and without an effective sensory trick (DYT-no-trick) (Experimental): Patients without an effective sensory trick will undergo a multimodal physiotherapy program for 6 weeks
  Interventions: Behavioral: Multimodal physiotherapy program
- Healthy subjects (No Intervention): Age- and sex-matched healthy subjects recruited to compare clinical and MRI characteristics at baseline.

INTERVENTIONS:
Behavioral: Multimodal physiotherapy program — Multimodal physiotherapy program of 6 weeks (3 times a week for 45 minutes), each session will include:
  * Soft tissue mobilization of inoculated muscles;
  * Stretching exercises of the inoculated muscles;
  * Strengthening of antagonist muscles;
  * Motor learning exercises (attentive strategies, feedback-based cervical active exercises).
  Exercises will be progressively difficult (increase of active ROM) according to clinical improvements.
  Arms: Patients with Cervical Dystonia and an effective sensory trick (DYT-trick); Patients with Cervical Dystonia and without an effective sensory trick (DYT-no-trick)

SUMMARY:
The primary aim of this study is to investigate improvements of dystonia severity in patients with cervical dystonia (CD) with (DYT-trick) and without sensory trick (DYT-no-trick) following 6 weeks of physiotherapy combined with botulinum toxin injection (BoNT).

The recruited patients will be divided into two groups according to the presence of an effective sensory trick (DYT trick and DYT no-trick groups).

The researchers analyzing clinical, neurophysiological and MRI data as well as the statistician will be blind about the allocation of subjects to the two groups. Considering the different clinical phenotypes of patients (DYT-trick and DYT-no-trick) clinical evaluators and physiotherapists cannot be blind.

All patients will perform the routinely BoNT injection and after 1 week they will start a multimodal physiotherapy program lasting 6 weeks, 3 times a week for 45 minutes each session. The physiotherapy treatment will include soft tissue mobilization of inoculated muscles, stretching exercises of the inoculated muscles, strengthening of antagonist muscles, and motor learning exercises (attentive strategies, feedback-based cervical active exercises). Exercises will be progressively difficult (increase of active range of motion -ROM) according to clinical improvements during the 6 weeks of treatment.

Clinical assessments will be performed at baseline (T0), after 6 weeks of treatment (W6) and before the next BoNT injection (about 12 weeks of follow-up, W12) to evaluate disease severity (TWSTRS), pain, active cervical range of motion, disability, quality of life and mood. Cervical movements during TWSTRS will be monitored using the Virtual Reality Rehabilitation System (VRRS), which includes the usage of magneto-inertial sensors to objectively assess joint positions and quality of movement. MRI evaluations will be performed at T0 and at W6 to investigate resting state functional Magnetic Resonance Imaging (fMRI) changes and fMRI changes of brain activation during the simulation and imagination of sensory trick.

SAI paradigm is obtained combing transcranial magnetic stimulation (TMS) with peripheral electrical stimulation techniques. It will be performed at baseline (before BoNT injection and physiotherapist training) and after week 6 of physiotherapist training.

A group of healthy subjects similar for age and sex to patients will be recruited to perform cognitive assessment and MRI at baseline.

ELIGIBILITY:
Inclusion Criteria fo patients with Cervical Dystonia:

* Adult onset idiopathic CD according to established diagnostic criteria (Albanese et al., Eur J Neur, 2011) with and without an effective sensory trick will be eligible for the study

Exclusion Criteria for all participants

* presence of fixed postures because of skeletal neck deformity;
* history of (other) systemic, neurologic, psychiatric diseases, head injury, cardiovascular events, and cerebrovascular alterations visible at an MRI scan;
* alcohol and/or psychotropic drugs abuse;
* contraindication to perform MRI scan (cardiac pace-maker or other types of cardiac catheters, splinters or metallic shards, metallic prosthesis not compatible with magnetic field generated by MRI, claustrophobia).

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 49 (Estimated)
Dates: Start 2019-04-13 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Toronto Western Spasmodic Rating Scale (TWSTRS) score | Baseline, after training (week 6) and 6 weeks after the end of training (week 12)
  Rating scale measuring severity, disability and pain associated with cervical dystonia (score 0-85, higher score = worse condition)

SECONDARY OUTCOMES:
Cervical range of motion | Baseline, after training (week 6) and 6 weeks after the end of training (week 12)
  Measure cervical active ROM (flexion, extension and lateral flexion) using electromagnetic sensors and the Virtual Reality Rehabilitation System (VRRS)
Cervical Dystonia Impact Scale (CDIP-58) score | Baseline, after training (week 6) and 6 weeks after the end of training (week 12)
  Questionnaire assessing the impact of cervical dystonia on activities of daily living, mood and health (score 0-100, higher score = higher impact)
Beck Depression inventory (BDI) score | Baseline, after training (week 6) and 6 weeks after the end of training (week 12)
  Evaluates depression (score 0-63, higher score = worse depressive symptoms)
Hamilton Anxiety Rating Scale (HAM-A) score | Baseline, after training (week 6) and 6 weeks after the end of training (week 12)
  Evaluates anxiety (score 0-56, higher score = worse anxiety symptoms)
Short-latency afferent inhibition (SAI) paradigm using transcranial magnetic stimulation (TMS) | Baseline, after training (week 6)
  TMS will be performed with a high power Magstim 200. A figure-of-eight Coil (70 mm external diameter) will be positioned over the hand area of the motor cortex. Motor evoked potentials (MEPs) will be recorded from first dorsal interosseous muscle (FDI) of the hand not performing the sensory trick. Resting motor threshold (RMT) will be determined starting below the expected threshold, with 5% stimulator output increments. RMT will be reported as percentage of maximum stimulator output (% MSO). To assess the SAI a conditioning electrical pulses will be applied through a bipolar electrode to the median nerve (not involved in sensory trick) at the wrist (cathode proximal). SAI will be randomly applied in two conditions: (A) at rest, with the patient's head positioned according to its dystonic pattern and (B) while patients will be performing the sensory trick
Brain functional changes during functional magnetic resonance imaging (MRI) task | Baseline, after training (week 6)
  A block design (ABAB) will be used, in which activation periods (A) alternated with resting-state periods (B). During activation periods (at the acoustic signal "go") DYT-trick patients will be asked to imagine their own effective sensory trick while DYT no-trick will imagine a simulation of sensory trick. Before scanning, participants will familiarize with the experimental condition.
Brain functional changes during functional magnetic resonance imaging (MRI) "conventional" resting state | Baseline, after training (week 6)
  Subjects will be instructed to remain motionless and to keep their eyes closed
Brain functional changes during functional magnetic resonance imaging (MRI) "sensory trick" resting state | Baseline, after training (week 6)
  Before scanning DYT subjects will be asked to execute (DYT-trick) or to simulate (DYT-no-trick) the sensory trick (i.e. slight touch on the cheek/chin) and to maintain it for the entire scanning. During scanning, DYT subjects will be instructed to remain motionless and to keep their eyes closed.

CONTACTS AND LOCATIONS:
Overall Officials: Massimo MF Filippi, MD, Principal Investigator — IRCCS Ospedale San Raffaele
Locations (1):
- IRCCS Ospedale San Raffaele, Milan, Italia, Italy